CLINICAL TRIAL: NCT04796792
Title: Ultrasound Technology to Fragment and Reposition Urinary Stones
Brief Title: Ultrasound to Facilitate Stone Passage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Indiana University (Other); VA Puget Sound Health Care System (U.S. Federal Agency); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jonathan Harper, MD, Associate Professor, School of Medicine, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00011687; 5P01DK043881-26 (NIH)
Record Dates: First submitted 2021-03-03; First posted 2021-03-15 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Urinary Stone; Urinary Calculi
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Intervention Model Description: Each phase represents a different population group. Phase 2a includes a randomized control component; the treatment and control groups are listed as separate arms with non-randomized allocation for consistency.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Phase I: Feasibility Treatment group (Experimental): Initial phase of the trial to demonstrate feasibility. All subjects undergo the investigational intervention.
  Interventions: Device: Burst Wave Lithotripsy (BWL) and Ultrasonic Propulsion (UP)
- Phase 2a: Treatment Group of a randomized control trial (Experimental): RCT phase of the trial to demonstrate superiority. All subjects undergo the investigational intervention.
  Interventions: Device: Burst Wave Lithotripsy (BWL) and Ultrasonic Propulsion (UP)
- Phase 2a: Control group of a randomized control trial (No Intervention): RCT phase of the trial to demonstrate superiority. All subjects are the concurrent Control to the Phase 2a Treatment group. Subjects receive no intervention.
- Phase 2b: Spinal Cord Injury Feasibility Study (Experimental): Feasbility study of the investigational intervention in subjects with spinal cord injury.
  Interventions: Device: Burst Wave Lithotripsy (BWL) and Ultrasonic Propulsion (UP)

INTERVENTIONS:
Device: Burst Wave Lithotripsy (BWL) and Ultrasonic Propulsion (UP) — Novel ultrasound technologies to facilitate passage of stones.This includes Burst Wave Lithotripsy (BWL), a technology to noninvasively fragment urinary calculi within the kidney and ureter, and ultrasonic propulsion, a technology to non-invasively reposition stones within the kidney and ureter. BWL uses short multi-cycle bursts of low amplitude ultrasound to induce stone fracture. This is in contrast to traditional extracorporeal shock wave lithotripsy (SWL), which employs a brief single compression/tensile cycle of high amplitude (shock) waves to achieve stone fracture. Ultrasonic propulsion uses long multi-cycle bursts of low amplitude ultrasound to move stones within the collecting system.
  Arms: Phase 2a: Treatment Group of a randomized control trial; Phase 2b: Spinal Cord Injury Feasibility Study; Phase I: Feasibility Treatment group

SUMMARY:
This is a prospective, open-label, multi-center study to test the clinical feasibility of facilitating stone passage by the combination of breaking and repositioning stones with ultrasound, without the need for anesthesia.

DETAILED DESCRIPTION:
This is a prospective, open-label, multi-center study to test the clinical feasibility of facilitating stone passage by the combination of breaking and repositioning stones with ultrasound, without the need for anesthesia.

Subjects will be included across three phases:

* Phase 1: 20 subjects to demonstrate initial feasibility
* Phase 2a: 100 subjects for a two-arm (50:50) randomized control trial (RCT)
* Phase 2b: 20 subjects to demonstrate feasibility in individuals with spinal cord injury (SCI)

This study has completed Phase 1. The study is currently recruiting for Phase 2b. Recruitment has not yet started for Phase 2a.

Up to 3 distinct targets may be treated per subject. The maximum total dose exposure is 30 minutes for one session. Subjects may return after at least 21 days and after all AEs have resolved for an additional session on the same side. Subjects may return after imaging follow-up for inclusion of their contralateral side.

ELIGIBILITY:
Inclusion Criteria:

* Individuals presenting with at least one kidney stone
* Stone with maximum dimension > 2 mm and ≤ 7 mm as determined by clinical imaging
* Individuals with SCI - (Phase 2b only)

Exclusion Criteria:

* Individuals under 18 years of age
* Individuals who are pregnant or who are trying to get pregnant
* Prisoners
* with cognitive impairment that would limit their ability to comprehend their role in consent or participation.
* Individuals who are unable to read or understand English
* Individuals who are unable or unwilling to participate in follow up activities
* Individuals who cannot be positioned for ultrasound imaging
* Individuals with uncorrected bleeding disorders or coagulopathies
* Individuals receiving anticoagulants and who are unable or not willing to temporarily cease the medication for the investigational procedure
* Individuals with a calcified abdominal aortic aneurysm or calcified renal artery aneurysm ipsilateral to the renal stone targeted by the investigational procedure
* Individuals with a solitary kidney
* Individuals with an uncorrected urinary tract obstruction
* Individuals with an untreated infection
* Individuals with a comorbidity risk which, at the discretion of the physician, would make the patient a poor candidate for the investigational procedure
* Individuals who have received two previous investigational procedures for the same stone target
* Individuals who have undergone the investigational procedure within the last 21 days or still have unresolved AEs from a previous investigational procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety - incidence of return healthcare visits. | Day of procedure to 14 months post-procedure
  Incidence of return health care visits associated with the device or procedure.
Effectiveness - stone comminution into fragments 2 mm or less. | Day of procedure to 4 months posts procedure
  Number of cases where the largest dimension of any residual stone in the study kidney is less than or equal to 2 mm.

SECONDARY OUTCOMES:
Safety - incidence of adverse events (AEs) | Day of procedure to 4 months posts procedure
  The incidence of all adverse events (AEs) associated with the device or procedure
Effectiveness - % residual stone volume | Day of procedure to 4 months posts procedure
  Residual stone volume relative to the initial stone volume
Effectiveness - need for further stone management | Day of procedure to 4 months posts procedure
  Incidence of new healthcare visits for further stone management
Effectiveness - Outcome from Wisconsin Stone Quality of Life questionnaire | Day of procedure to 14 months posts procedure
  Quality of life, evaluated by the comparison of Wisconsin Stone Quality of Life (WISQOL) questionnaire scores before and after the investigational procedure. The questionnaire consists of a series of questions to evaluate the symptomatic and functional impact of the stones on a scale of 1 to 5, where a lower score indicates a greater impact. https://urology.wisc.edu/research/wisqol/.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Harper, MD, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - Indiana University Health - North Hospital, Carmel, Indiana
  - VA Puget Sound Health Care System, Seattle, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] May PC, Kreider W, Maxwell AD, Wang YN, Cunitz BW, Blomgren PM, Johnson CD, Park JSH, Bailey MR, Lee D, Harper JD, Sorensen MD. Detection and Evaluation of Renal Injury in Burst Wave Lithotripsy Using Ultrasound and Magnetic Resonance Imaging. J Endourol. 2017 Aug;31(8):786-792. doi: 10.1089/end.2017.0202. Epub 2017 Jun 16. PMID 28521550
- [Background] Maxwell AD, Cunitz BW, Kreider W, Sapozhnikov OA, Hsi RS, Harper JD, Bailey MR, Sorensen MD. Fragmentation of urinary calculi in vitro by burst wave lithotripsy. J Urol. 2015 Jan;193(1):338-44. doi: 10.1016/j.juro.2014.08.009. Epub 2014 Aug 9. PMID 25111910
- [Background] Harper JD, Metzler I, Hall MK, Chen TT, Maxwell AD, Cunitz BW, Dunmire B, Thiel J, Williams JC, Bailey MR, Sorensen MD. First In-Human Burst Wave Lithotripsy for Kidney Stone Comminution: Initial Two Case Studies. J Endourol. 2021 Apr;35(4):506-511. doi: 10.1089/end.2020.0725. Epub 2020 Nov 5. PMID 32940089
- [Background] Ramesh S, Chen TT, Maxwell AD, Cunitz BW, Dunmire B, Thiel J, Williams JC, Gardner A, Liu Z, Metzler I, Harper JD, Sorensen MD, Bailey MR. In Vitro Evaluation of Urinary Stone Comminution with a Clinical Burst Wave Lithotripsy System. J Endourol. 2020 Nov;34(11):1167-1173. doi: 10.1089/end.2019.0873. Epub 2020 Mar 20. PMID 32103689
- [Background] Dai JC, Sorensen MD, Chang HC, Samson PC, Dunmire B, Cunitz BW, Thiel J, Liu Z, Bailey MR, Harper JD. Quantitative Assessment of Effectiveness of Ultrasonic Propulsion of Kidney Stones. J Endourol. 2019 Oct;33(10):850-857. doi: 10.1089/end.2019.0340. Epub 2019 Sep 25. PMID 31333058
- [Background] Maxwell AD, Wang YN, Kreider W, Cunitz BW, Starr F, Lee D, Nazari Y, Williams JC Jr, Bailey MR, Sorensen MD. Evaluation of Renal Stone Comminution and Injury by Burst Wave Lithotripsy in a Pig Model. J Endourol. 2019 Oct;33(10):787-792. doi: 10.1089/end.2018.0886. Epub 2019 May 27. PMID 31016998
- [Background] Harper JD, Cunitz BW, Dunmire B, Lee FC, Sorensen MD, Hsi RS, Thiel J, Wessells H, Lingeman JE, Bailey MR. First in Human Clinical Trial of Ultrasonic Propulsion of Kidney Stones. J Urol. 2016 Apr;195(4 Pt 1):956-64. doi: 10.1016/j.juro.2015.10.131. Epub 2015 Oct 30. PMID 26521719
- [Background] Harper JD, Lingeman JE, Sweet RM, Metzler IS, Sunaryo PL, Williams JC Jr, Maxwell AD, Thiel J, Cunitz BW, Dunmire B, Bailey MR, Sorensen MD. Fragmentation of Stones by Burst Wave Lithotripsy in the First 19 Humans. J Urol. 2022 May;207(5):1067-1076. doi: 10.1097/JU.0000000000002446. Epub 2022 Mar 21. PMID 35311351
- [Background] Hall MK, Thiel J, Dunmire B, Samson PC, Kessler R, Sunaryo P, Sweet RM, Metzler IS, Chang HC, Gunn M, Dighe M, Anderson L, Popchoi C, Managuli R, Cunitz BW, Burke BH, Ding L, Gutierrez B, Liu Z, Sorensen MD, Wessells H, Bailey MR, Harper JD. First Series Using Ultrasonic Propulsion and Burst Wave Lithotripsy to Treat Ureteral Stones. J Urol. 2022 Nov;208(5):1075-1082. doi: 10.1097/JU.0000000000002864. Epub 2022 Nov 1. PMID 36205340
- [Background] Sorensen MD, Dunmire B, Thiel J, Cunitz BW, Burke BH, Levchak BJ, Popchoi C, Holmes AE, Kucewicz JC, Hall MK, Dighe M, Dai JC, Cormack FC, Liu Z, Bailey MR, Porter MP, Harper JD. Randomized Controlled Trial of Ultrasonic Propulsion-Facilitated Clearance of Residual Kidney Stone Fragments vs Observation. J Urol. 2024 Dec;212(6):811-820. doi: 10.1097/JU.0000000000004186. Epub 2024 Aug 15. PMID 39146526
- [Background] Shelton TM, Connors BA, Rivera ME, Lingeman JE, Bailey MR, Williams JC Jr. No Injury Observed in Kidneys Treated with Burst Wave Lithotripsy in Therapeutically Anticoagulated Pigs. J Endourol. 2025 Aug;39(8):804-807. doi: 10.1089/end.2024.0466. Epub 2025 Jan 16. PMID 39819022
- [Result] Harper JD, Dunmire B, Thiel J, Burke BH, Wang YN, Totten S, Kucewicz JC, Maxwell AD, Hall MK, Holmes AE, Popchoi C, Lingeman JE, Desai AC, Sweet RM, Dighe M, Levchak BJ, Yang CC, Bailey MR, Sorensen MD. Facilitated Clearance of Small, Asymptomatic Renal Stones With Burst Wave Lithotripsy and Ultrasonic Propulsion. J Urol. 2025 Jul;214(1):41-47. doi: 10.1097/JU.0000000000004533. Epub 2025 Mar 17. PMID 40096677
- See also: Sponsor website — http://www.apl.washington.edu/project/project.php?id=bwl